CLINICAL TRIAL: NCT02775578
Title: Study of Serum Level of Heart Failure Related Biomarkers and Optimization Strategy of Coronary Revascularization in Patients With Multivessel Lesions Combined Heart Failure
Brief Title: Optimizing Strategy of Coronary Revascularization in Patients With Multivessel Lesions Combined Heart Failure
Acronym: OSCRM-HF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Zhang Qi, MD, Chief docter, Shanghai Jiao Tong University School of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RJH20160405
Record Dates: First submitted 2016-04-26; First posted 2016-05-17 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Heart Failure Due to Coronary Artery Disease
Keywords: heart failure; coronary artery disease; biomarkers; Percutaneous Coronary Intervention, PCI; Coronary Artery Bypass Grafting, CABG
MeSH Terms: conditions — Heart Failure; Coronary Artery Disease | interventions — Coronary Artery Bypass; Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Coronary Artery Bypass Grafting (Experimental): Using coronary artery bypass grafting surgery as the coronary revascularization therapy for patients enrolled.
  Interventions: Procedure: Coronary Artery Bypass Grafting
- Percutaneous Coronary Intervention (Experimental): Using percutaneous coronary intervention as the coronary revascularization therapy for patients enrolled.
  Interventions: Procedure: Percutaneous Coronary Intervention
- Hybrid Coronary Revascularization (Experimental): Patients enrolled will take coronary artery bypass grafting surgery at first, then treated with percutaneous coronary intervention.
  Interventions: Procedure: Hybrid Coronary Revascularization

INTERVENTIONS:
Procedure: Coronary Artery Bypass Grafting — Using coronary artery bypass grafting surgery as the coronary revascularization therapy for patients enrolled.
  Arms: Coronary Artery Bypass Grafting
Procedure: Percutaneous Coronary Intervention — Using percutaneous coronary intervention as the coronary revascularization therapy for patients enrolled.
  Arms: Percutaneous Coronary Intervention
Procedure: Hybrid Coronary Revascularization — Patients enrolled will take coronary artery bypass grafting surgery at first, then treated with percutaneous coronary intervention.
  Arms: Hybrid Coronary Revascularization

SUMMARY:
As the end stage of almost all cardiovascular diseases, heart failure has become an increasingly common cause of cardiovascular morbidity and mortality worldwide. In China, coronary artery disease (CAD) has become the main cause of heart failure in recent years. CAD combining with heart failure usually predicts poor outcome, with coronary revascularization the most universally used therapy. However, the difference of several types of such therapy has less well been compared.

Thus, the study mainly aims to compare different types of coronary revascularization therapies such as Percutaneous Coronary Intervention (PCI),Coronary Artery Bypass Grafting (CABG) as well as Hybrid Coronary Revascularization (HCR), and also make the optimization strategy especially in patients with heart failure.

The study also aims to investigate whether disease progression in patients with chronic heart failure (CHF) can be assessed by new biomarkers and determine their diagnostic and prognostic value, relating several cardiac functional parameters to clinical outcome.

DETAILED DESCRIPTION:
STUDY DESIGN This is a single center prospective study mainly designed to compare different types of coronary revascularization therapies in patients with severe coronary artery disease combining heart failure. We will collect the data at baseline before the therapy, as well as 30 days, 6 months and 12 months after surgery. Using follow-up visits along with effective exams such as echocardiography, cardiopulmonary function mensuration and tests of serum markers, we will principally make a comparison of both primary and secondary outcomes, also quality of life among patients in these three groups.

STUDY POPULATION About 525 patients who are diagnosed with severe CAD and HF will be enrolled. Severe CAD is defined as at least 2 vessel disease with each ≥50% narrowing of the luminal diameter shown by coronary angiography, including LAD. Those enrolled also has reduced cardiac systolic function (LVEF≤50%).

STUDY DURATION It will take about 2 years to finish all follow-up visits with each patient at least 12 months after surgery.

STUDY PROCESS The statistical analysis will include all the materials of each patient in every follow-up visit. We will describe basic characteristics and test parameters of every visit, comparing those in PCI, CABG and HCR group, to further investigate the prognostic influence of each therapeutic method.

Data analysis will be processed by SPSS. All the analysis will be used by the 2-side test with 95% confidence interval, showing statistical significance if 2-side p value is less than 0.05. The study will finally report primary and secondary outcomes, as well as changes of several important parameters.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* with at least 2 lesion vessels defined as ≥50% narrowing of the luminal diameter as shown by coronary angiography, including LAD
* LVEF≤50% as shown in echocardiography

Exclusion Criteria:

* with other severe diseases combined and will be alive for less than 12 months
* combining valvular heart disease
* pregnant or lactating women
* during the acute phase of ST-elevation acute myocardial infarction
* with severe renal dysfunction requiring dialysis to cure
* hard to participate in the investigation or accept the follow-up visits
* those who have already taken PCI treatment before
* with other diseases which need to be treated by surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 525 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
main adverse cardiovascular and cerebrovascular events, MACCE | 12 months
  MACCE includes all-cause mortality, cardiovascular mortality, nonfatal myocardial infarction, nonfatal stroke, target lesion revascularization and HF rehospitalization

SECONDARY OUTCOMES:
all-cause mortality | 12 months
cardiovascular mortality | 12 months
new myocardial infarction | 12 months
new stroke | 12 months
heart failure rehospitalization | 12 months
quality of life | 12 months
  described in quality of life score
decline of left ventricular ejection fraction | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided